CLINICAL TRIAL: NCT07252648
Title: Effect of Peri-Operative Music Therapy on Anxiety, Pain Catastrophising, and Pain in Chronic Pain Patients Undergoing Interventional Pain Procedures - A Randomised Controlled Trial
Brief Title: Music Therapy to Reduce Anxiety and Pain in Chronic Pain Patients During Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025-1781
Record Dates: First submitted 2025-11-18; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain; Anxiety; Music Therapy; Pain Perception; Pain Catastrophizing
Keywords: Pain Catastrophizing; Music Therapy; Anxiety; Chronic Pain
MeSH Terms: conditions — Chronic Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): Participants will listen to self-selected music before, during, and after the interventional pain procedure via headphones. Bluetooth speakers will be used during the procedure to facilitate communication with the healthcare team.
  Interventions: Behavioral: Music Therapy
- Standard Care (No Intervention): Participants will receive routine peri-procedural care without music therapy.

INTERVENTIONS:
Behavioral: Music Therapy — This intervention consists of perioperative music therapy for patients with chronic pain undergoing interventional pain procedures in the ambulatory setting. Participants in the intervention group will listen to self-selected music for approximately 30 minutes before, during the procedure, and 30 minutes after their procedure. Music will be delivered via headphones pre- and post-procedure and via a Bluetooth speaker during the procedure to facilitate communication with the procedural team.
  Arms: Music Therapy

SUMMARY:
This study aims to find out whether listening to music before, during, and after pain procedures can help reduce anxiety, pain catastrophising, and acute pain in patients with chronic pain. Music therapy may provide a simple, safe, and non-drug way to help patients relax and feel more comfortable.

In this study, adult patients with chronic pain who are scheduled for interventional pain procedures at Singapore General Hospital will be randomly assigned to one of two groups. One group will listen to self-selected music through headphones and speakers before, during, and after the procedure. The other group will receive standard care without music.

Researchers will measure anxiety, pain catastrophising, and pain levels before and after the procedure using validated questionnaires. The main outcome will be the level of anxiety after the procedure. Other outcomes include pain catastrophising scores, pain scores during local anaesthetic injection, and overall patient satisfaction.

This study will help determine if music therapy can be routinely used to improve comfort and emotional well-being for patients undergoing interventional pain procedures.

DETAILED DESCRIPTION:
This is a single-centre, randomised controlled trial conducted at the Singapore General Hospital Pain Management Centre. The study investigates whether peri-operative music therapy can reduce anxiety, pain catastrophising, and pain in patients with chronic pain undergoing interventional pain procedures in the ambulatory setting.

A total of 110 adult participants (aged 21 years and above) with chronic pain lasting at least 3 months and scheduled for interventional pain procedures will be enrolled. Participants will be randomised in a 1:1 ratio to either the music therapy group or the control group using a computer-generated block randomisation sequence with sealed opaque envelopes.

Intervention group: Participants will listen to self-selected music from curated playlists (including soothing, meditative, multilingual, and instrumental tracks) before, during, and after the procedure. Music will be played for 30 minutes pre-procedure via headphones, continued intra-procedurally via Bluetooth speaker to maintain communication, and resumed for 30 minutes post-procedure via headphones.

Control group: Participants will receive standard peri-procedural care without music exposure.

Due to the nature of the intervention, blinding of participants and proceduralists is not feasible. However, outcome assessors and statisticians will remain blinded to group allocation.

The primary endpoint is postoperative anxiety measured using the Visual Analogue Scale for Anxiety (VAS-A) and the Hospital Anxiety and Depression Scale (HADS). Secondary endpoints include pain catastrophising scores (Pain Catastrophising Scale, PCS), procedural pain (Numerical Rating Scale, NRS), and patient satisfaction scores.

Data will be collected pre-procedure and immediately post-procedure. Baseline demographics, analgesic/sedative use, and intra-procedural variables (e.g., duration, complications, and rescue medication use) will also be recorded. Statistical analysis will compare mean differences between groups using independent t-tests for continuous variables and chi-square tests for categorical variables, with significance set at p < 0.05.

The study is classified as minimal risk, involving a non-invasive behavioural intervention. No Data Monitoring Committee has been appointed. Oversight will be provided by the Principal Investigator and study mentor, with periodic internal data reviews.

This trial aims to provide evidence for a simple, low-cost, and patient-centred intervention that could enhance peri-procedural comfort and reduce psychological distress in chronic pain patients undergoing day surgery procedures.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥21years
* chronic pain ≥3 months
* scheduled for interventional pain procedures

Exclusion Criteria:

* presence of hearing impairment
* lack of capacity to consent
* non-interventional pain procedures, e.g. lignocaine infusion, ketamine infusion
* pregnant women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative Anxiety (Visual Analogue Scale) | Scores will be recorded before the procedure (baseline) and post-procedure within 30 minutes.
  Postoperative anxiety will be assessed using the Visual Analogue Scale for Anxiety, a 10-cm scale ranging from 0 (not anxious at all) to 10 (extremely anxious).

SECONDARY OUTCOMES:
Pain Catastrophising Score | This will be measured before the procedure (baseline) and post-procedure within 30 minutes.
  Pain catastrophising will be assessed using the Pain Catastrophising Scale, which measures rumination, magnification, and helplessness related to pain. Each item is rated from 0 (not at all) to 4 (all the time), with total scores ranging from 0 to 52.
Postoperative Anxiety (State-Trait Anxiety Inventory Short Form) | This will be measured at baseline (pre-procedure) and post-procedure (within 30 minutes of completion).
  State anxiety will be measured using the State-Trait Anxiety Inventory - Short Form (STAI-SF), a validated questionnaire assessing transient anxiety related to specific situations. Each item is rated on a 4-point scale, and total scores range from 20 to 80, with higher scores indicating greater anxiety.
Postoperative Pain Score | Participants will rate their pain after the procedure in the recovery area (within 30 minutes).
  Pain intensity will be assessed using an 11-point Numerical Rating Scale, where 0 = "no pain" and 10 = "worst pain imaginable."
Patient Satisfaction | Within 30 minutes of the procedure.
  Patient satisfaction will be assessed after the procedure using a 5-point Likert scale (1 = Very satisfied, 2 = Satisfied, 3 = Neutral, 4 = Dissatisfied, 5 = Very dissatisfied). Participants in both groups will rate their overall satisfaction with their perioperative experience.

OTHER OUTCOMES:
Patient Music Preferences | Post-procedure within 30 minutes.
  The music genres that participants listened to as part of the music therapy will recorded for participants in the music therapy group. Data will be presented descriptively for each category, and to explore associations between music genre and anxiety or pain outcomes.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li G, Yu L, Yang Y, Deng J, Shao L, Zeng C. Effects of Perioperative Music Therapy on Patients with Postoperative Pain and Anxiety: A Systematic Review and Meta-Analysis. J Integr Complement Med. 2024 Jan;30(1):37-46. doi: 10.1089/jicm.2022.0803. Epub 2023 Aug 30. PMID 37646752
- [Background] Goel SK, Kim V, Kearns J, Sabo D, Zoeller L, Conboy C, Kelm N, Jackovich AE, Chelly JE. Music-Based Therapy for the Treatment of Perioperative Anxiety and Pain-A Randomized, Prospective Clinical Trial. J Clin Med. 2024 Oct 15;13(20):6139. doi: 10.3390/jcm13206139. PMID 39458090
- [Background] Kakde A, Lim MJ, Shen H, Tan HS, Tan CW, Sultana R, Sng BL. Effect of music listening on perioperative anxiety, acute pain and pain catastrophizing in women undergoing elective cesarean delivery: a randomized controlled trial. BMC Anesthesiol. 2023 Apr 3;23(1):109. doi: 10.1186/s12871-023-02060-w. PMID 37013499